CLINICAL TRIAL: NCT05749744
Title: Effects of Cardiac Telerehabilitation During COVID-19 on Cardiorespiratory Capacities in Coronary Artery Disease Patients.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1022021/CHUSTE
Record Dates: First submitted 2023-02-27; First posted 2023-03-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Disease
Keywords: cardiac telerehabilitation; acute coronary syndrome; rehabilitation therapeutic; rehabilitation sessions; cardiorespiratory functions
MeSH Terms: conditions — Heart Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home-based cardiac telerehabilitation (interventional group): Patients followed the cardiac rehabilitation program at home.
  Interventions: Other: cardiac telerehabilitation program by videoconference
- Traditional centre-based cardiac rehabilitation (control group): Patients participates in the cardiac rehabilitation program in hospital.

INTERVENTIONS:
Other: cardiac telerehabilitation program by videoconference — * A video conference interview with an Adapted Physical Activity (APA) teacher before starting physical training
  * Exercise training for 3 weeks via distance coaching
  * Therapeutic patient education (TPE) workshops conducted remotely with 1 workshop per week.
  * Medical follow-up via teleconsultation
  * Psychological and/or dietetic follow-up if necessary.
  * Final assessment at 1 month with evaluation of aerobic metabolism, functional evaluation and final shared educational assessment (BEP).
  * Appointment with an association "Cœur et Santé" and "Sport-Santé 42" or setting up of an individual physical activity
  Groups: Home-based cardiac telerehabilitation (interventional group)

SUMMARY:
After an acute coronary syndrome, an adapted cardiac rehabilitation program is necessary to restore or increase physical capacities and decrease cardiovascular risk. This multidisciplinary care combines physical training sessions and therapeutic education workshops.

The COVID-19 pandemic imposed restrictions such as the closure of rehabilitation centres. To remedy this problem, one solution was to adapt the existing program to a remote cardiac telerehabilitation, i.e., medical and paramedical supervision of rehabilitation sessions and therapeutic patient education meetings via digital tools. Recent studies have shown that it was a safe (no reported adverse effects), effective (similar gains in peak oxygen consumption compared to traditional cardiac rehabilitation and patient-adherence alternative.

DETAILED DESCRIPTION:
The hypothesis of this study is that telerehabilitation was more effective on cardiorespiratory functions.

ELIGIBILITY:
Inclusion Criteria:

Both groups:

* Acute Coronary Syndrome treated in the last 6 months
* Medical revascularization (angioplasty ± stenting) or surgical (coronary artery bypass)

For Telerehabilitation group:

* Internet connexion (computer or digital tablet)
* Equipped with an exercise bike

Exclusion Criteria:

Both groups:

* Pulmonary hypertension
* Aortic pathway anomaly
* Uncontrolled ventricular rhythm disorders

For Telerehabilitation group:

* Important muscular deconditioning
* Patient requiring medical supervision in institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Acute Coronary Syndrome treated in the last 6 months will be included.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline oxygen (VO2) (ml/min/kg) at the first ventilatory threshold (VT1) at 2 months | Months: 0, 2
  Variation of oxygen (VO2) (ml/min/kg) at the first ventilatory threshold (VT1) during a cardio-pulmonary exercise test (CPET) before and after 15 training sessions performed

SECONDARY OUTCOMES:
oxygen (VO2) peak | Months: 0, 2
  Variation of oxygen (VO2) peak before and after 15 training sessions performed
maximum power workload | Months: 0, 2
  Variation of maximum power workload before and after 15 training sessions performed
power at the first ventilatory threshold (VT1) | Months: 0, 2
  Variation of power at the first ventilatory threshold (VT1) before and after 15 training sessions performed
maximum heart rate | Months: 0, 2
  Variation of maximum heart rate before and after 15 training sessions performed.
recovery heart rate | Months: 0, 2
  Variation of recovery heart rate before and after 15 training sessions performed.
obstructive ventilatory disorder | Months: 0, 2
  Variation of obstructive ventilatory disorder before and after 15 training sessions performed.
autonomic nervous system | Months: 0, 2
  Variation of autonomic nervous system before and after 15 training sessions performed.
muscular strength | Months: 0, 2
  Variation of muscular strength before and after 15 training sessions performed.
muscular endurance | Months: 0, 2
  Variation of muscular endurance before and after 15 training sessions performed.

CONTACTS AND LOCATIONS:
Overall Officials: David Hupin, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No